CLINICAL TRIAL: NCT06447480
Title: Randomized Clinical Trial to Compare Oral Isotretinoin to Standard of Care in Moderate Acne Skin of Color Patients: ETHNIC Study
Brief Title: Clinical Trial to Compare Oral Isotretinoin to Standard of Care in Moderate Acne Skin of Color Patients
Acronym: ETHNIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-APN-02
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; Floderm topical cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug group (Experimental): Patients will be followed every month for 6 months in the group isotretinoin. Patients will start at the dose of 0.5 mg/kg/d. If tolerance is poor, the dose could be decrease to 0.25mg/d. After 3 months, following the recommendations the dose could be increase up to 1mg/kg/d depending on the efficacy.
  Interventions: Drug: ISOtretinoin 5 MG
- Doxycycline (Active Comparator): Patients will be followed at 3 and 6 months in the group "standard of care". They will be prescribed topical tretinoin or adapalene once daily (every other day if irritation) with doxycycline or lymecycline 100 mg/d.
  Interventions: Drug: Topical cream

INTERVENTIONS:
Drug: ISOtretinoin 5 MG — The dose is usually of 0.5 mg/kg/d. If tolerance is poor, the dose of isotretinoin can be decreased to 0.25 mg/kg/d.
  After 3 months of treatment, a clinical evaluation is performed. The dose of isotretinoin can be increased up to 1 mg/kg/d depending on the efficacy (ECLA graded as moderated or severe) and tolerance. A total cumulative dose between 120 to 150 mg/kg is recommended.
  Arms: Drug group
Drug: Topical cream — Topical retinoic acid (Effederm®) or adapalene cream (Differine®), associated during the 3 first months with doxycycline or lymecycline 100 mg/d. After 3 months, the efficacy is assessed. If acne improved, oral antibiotics are stopped and only the topical treatment is continued. If the ECLA is graded as moderated or severe, isotretinoin should be introduced.
  Arms: Doxycycline

SUMMARY:
In Dermatology, assessment of people of color remains underrepresented in RCTs (<10%) and guidelines. Acne affects around 9% of the population worldwide and negatively affects quality of life and self-esteem with anxiety, suicidal ideation and physical scarring. Main lesions associate comedons, inflammatory papules and pustules which grading of severity allows decision-making, e.g., topicals in mild acne and isotretinoin in severe acne. In darker skin type patients, i.e., Fitzpatrick phototypes IV-VI, acne-related pigmentation (ARP) occurs in 65% of cases which reflects either per- or post-inflammatory hyperpigmentation. Whatever is the mechanism, ARP (number, size, importance of dyschromia) impacts the quality of life in such patients. In moderate acne, treatment is based on oral antibiotics for 3 months, i.e., doxycycline or lymecycline, with topical treatment like tretinoin targeting comedons (and potentially ARP). However, oral antibiotics first-line were developed in white skin patients only and never showed its efficacy in ARP. Moreover, doxycycline could be associated with new-onset hyperpigmentation in acne patients. Isotretinoin -acting on the sebaceous gland and therefore the most effective drug in acne- is only prescribed after failure of antibiotics according to the guidelines.The main objective: To assess the superiority at M6 of a treatment of moderate facial acne in skin of color patients with oral isotretinoin in first line compared to the current standard of care on the severity of ARP.Multicenter randomized controlled trial - open study. The number of subjects required for the trial = 420

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 13 and 30-year-old
* Skin type IV, V and VI according to Fitzpatrick skin types
* Moderate acne as defined by the French Society of Dermatology recommendations based on ECLA grading https://document.sfdermato.org/groupe/centre-de-preuves/label-recommandations-acne-post-college.pdf)
* Patients must have a cell phone able to take selfies pictures with a minimum definition of 5Mb.
* Signed informed consent
* Affiliation to French social coverage.

Exclusion Criteria:

* Mild and severe acne (ECLA grading : French recommendations) (https://document.sfdermato.org/groupe/centre-de-preuves/label-recommandations-acne-post-college.pdf)
* Past cure of oral isotretinoin
* Past cure of systemic antibiotics for acne in the last 6 months
* Phototype I-III patients
* Abnormal hemogram, liver enzyme, cholesterol, triglycerides at baseline
* Pregnancy: female patient of childbearing potential will undergo a pregnancy test (plasmatic β-hCG)
* Breast-feeding patients
* Refusal of effective contraception for women
* Contra-indications to oral isotretinoin, doxycycline, lymecycline, topical adapalene/tretinoin
* Vulnerable people: adult under guardianship or deprived of freedom

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of score acne-related pigmentation | at 6 months
  To assess the superiority after 6 months of a first line oral isotretinoin treatment of moderate facial acne in skin of color patients compared to the current standard of care on the severity of ARP.

SECONDARY OUTCOMES:
Quality of life of patient | at 6 months
  Quality of life will be evaluated with the Acne-specific Quality of Life questionnaire (Acne-QoL)
Number of adverse events | during 6 months
  A special focus on scars will be performed using an Investigator Global Assessment score (0 no scar, 1 mild scarring, 2 moderate, 3 severe) over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (16):
- France (15):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes
  - CHU de Bordeaux, Bordeaux, Aquitaine
  - CHU de Nantes, Nantes, Loire-Atlantique
  - chu de Rouen, Rouen, Seine-maritime
  - Cabinet de dermatologie St Maxime, Sainte-Maxime, Var
  - CH D'argenteuil, Argenteuil
  - Cabinet Dermatologique Brest 1, Brest
  - Cabinet Dermatologique Brest 2, Brest
  - Cabinet dermatologique Cenon, Cenon
  - Cabinet dermatologique gradignan, Gradignan
  - CHU de la réunion, La Réunion
  - Cabinet dermatologique privé, Paris
  - CH Avicenne - APHP, Paris
  - Hôpital Béclére, Paris
  - APHP, Paris, Île-de-France Region
- CH de Cayenne 3 Avenue Alexis Blaise, BP6006, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided